CLINICAL TRIAL: NCT05388045
Title: Piloting a Patient-Reported Outcome Measure for Opioid Use Disorder Recovery in a Clinical Setting
Acronym: RecoveryPROM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Brandeis University (Other)
Collaborators: Stanley Street Treatment and Resources (SSTAR) (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sharon Reif, Professor, Brandeis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19123R; R61DA049263 (NIH)
Record Dates: First submitted 2022-05-13; First posted 2022-05-24 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Substance Use Disorders; Opioid Use Disorder
Keywords: Patient reported outcome measure; Recovery; Measure development
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Intervention Model Description: No randomization is involved, with all eligible patients invited to participate.
Masking Description: The intervention is not blinded to patients, clinicians, or investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recovery PROM (Experimental): All study participants will complete the Recovery PROM instrument.
  Interventions: Other: Patient Reported Outcome Measure

INTERVENTIONS:
Other: Patient Reported Outcome Measure — A Recovery Patient-Reported Outcome Measure (PROM, 19 items and 2 questions for each item, collected via online survey) will be completed by eligible patients at baseline and again at months 3 and 6. The initial Recovery PROM will be shared with the clinician, at the visit most closely scheduled following the baseline visit, for review and discussion with the patient. At the 3- and 6-month visits, the clinician will be asked to re-review and compare the earlier Recovery PROM(s) as well as the current Recovery PROM. The clinician is encouraged to use the PROM results during interim clinical visits with the patient. Efforts will be made to contemporaneously track how often the PROM is discussed in clinical sessions conducted during the 6 months.

SUMMARY:
Performance measure can improve quality of care at the patient, provider, and systems level of care, and patient-reported outcome measures bring a needed patient-centered focus. Recovery has been difficult to measure for people with substance use disorders, and is more challenging in the context of opioid use disorders (OUD) and treatment medications. This study will examine a recovery patient-reported outcome measure to determine if patients and clinicians find it useful and acceptable in the clinical context, and if it leads to improved outcomes.

DETAILED DESCRIPTION:
The pilot clinical trial will test the newly developed Recovery Patient-Reported Outcome Measure ("Recovery PROM") and approach with patients and clinicians in an office-based opioid medication treatment program (known as office-based opioid treatment (OBOT), medication-assisted treatment (MAT) or medications for OUD (MOUD)), in the specific context of buprenorphine treatment.

Aims

This is a pilot study to assess the feasibility of implementing the Recovery PROM into the workflow of a clinical setting, assess its initial effectiveness, and evaluate its value to patients and clinicians. The aims are as follows:

1. Work with a clinical partner to assess and refine the draft Recovery PROM, and examine feasibility and implementation (e.g., workflow, data transfer issues) related to its use in a clinical setting.
2. Determine initial effectiveness of the Recovery PROM for improving patient outcomes (self-efficacy, health-related quality of life, patient-provider relationship, social determinants of health, substance use) and facilitating self-directed care and patient-centered shared decision-making.
3. Evaluate and update (if needed) the Recovery PROM in terms of recovery while on OUD medication treatment, patient characteristics, and clinical workflow.

Hypotheses Although this pilot study is primarily for information gathering, and ultimately refinement of the Recovery PROM and approach, the study has two broad hypotheses.

H1. Patients and clinicians will find the Recovery PROM to be a useful tool for patient recovery.

H2. Patient self-efficacy, shared decision-making, patient-provider relationship, and health-related quality of life will improve and substance use will decrease with the use of the Recovery PROM.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Taking buprenorphine for OUD treatment, in current episode of care at clinical partner site, for at least 6 weeks but less than 3 years.
* Able and willing to provide informed consent.
* Able to read English, to provide informed consent and complete study instruments.
* Able to use a smart phone to complete study instruments [phones with data plan will be provided for those without].

Exclusion Criteria:

• Patients who do not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in reported health related quality of life (4-point scale), assessed via CDC HRQOL questionnaire | 3 months after baseline, 6 months after baseline
  Centers for Disease Control & Prevention (CDC) Health Related Quality of Life (HRQOL) questionnaire, single item ranging from excellent (score=1) to poor (score=5).
Change in number of days mental/physical health were not good (in past 30 days), assessed via CDC HRQOL questionnaire. | 3 months after baseline, 6 months after baseline
  CDC Health Related Quality of Life (HRQOL) questionnaire, separate items for mental and physical health, single item measuring the number of days out of 30, where 0 is no days (better) and 30 is daily (worse).
Change in reported self-efficacy for managing chronic conditions, assessed via PROMIS Self-Efficacy measure | 3 months after baseline, 6 months after baseline
  Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy scale, a series of 10 questions each on a 5-point scale, ranging from not at all confident (score=1) to very confident (score=5).
Change in patient-clinician alliance, assessed via WAI-SR | 3 months after baseline, 6 months after baseline
  Working Alliance Inventory-Short Revised (WAI-SR): Patient-clinician alliance for tasks and goals of treatment, and effective relationship. This scale is a series of 12 items, with responses ranging from seldom (score=1) to always (score=5).

SECONDARY OUTCOMES:
Social determinants of health, assessed via PRAPARE | 3 months after baseline, 6 months after baseline
  Protocol for Responding to and Assessing Patient Assets, Risks, and Experiences (PRAPARE). The prepare is a series of independent questions related to social determinants of health; it is not scored.
Substance use past 30 days, assessed via modified ASI Alcohol and Drug module | 3 months after baseline, 6 months after baseline
  Modified Alcohol and Drug module of the Addiction Severity Index (ASI). The ASI asks how many days in the past 30 each substance was used, where 0 is no use (better) and 30 days is daily use (worse).

OTHER OUTCOMES:
Satisfaction with Recovery PROM | 6 months after baseline
  Self-developed questions. These are independent questions. Each is scored on a scale of 1 to 5, where 1 is the best outcome (e.g., extremely satisfied) and 5 is the worst outcome (e.g., extremely unsatisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Reif, PhD, Principal Investigator — Brandeis University; Constance M Horgan, ScD, Principal Investigator — Brandeis University
Locations (1):
- Stanley Street Resources and Treatment, Fall River, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okrant E, Reif S, Horgan CM. Development of an addiction recovery patient-reported outcome measure: Response to Addiction Recovery (R2AR). Subst Abuse Treat Prev Policy. 2023 Sep 1;18(1):52. doi: 10.1186/s13011-023-00560-z. PMID 37658373